CLINICAL TRIAL: NCT00346112
Title: Rehabilitation, Quality of Life, and Exercise Tolerance in Internal Cardioverter-Defibrillator-patients, RELAX-ICD Trial
Brief Title: Rehabilitation, Quality of Life, and Exercise Tolerance in Patients With an ICD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P-KARE-01
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Heart Patients After ICD Implantation
Keywords: ICD; distress; anxiety; quality-of-life
MeSH Terms: conditions — Anxiety Disorders

INTERVENTIONS:
Procedure: psycho-educational

SUMMARY:
RELAX-ICD Trial/Research Study; Quality of Life/Protocol No.P-KARE-01: A 3-month outpatient rehabilitation therapy and psychological counselling including informative talks with conventional therapy, by a cardiologist or general practitioner after implantation of an internal cardioverter defibrillator (ICD) in adult patients, whereby the effects of three different strategies are compared. Study hypothesis: the rehabilitation programme will be beneficial in the management of any psychological problems possibly as a result from the intervention, and will help to overcome anxiety, and contribute to improved quality of life.

DETAILED DESCRIPTION:
University Hospital Inselspital Berne,Switzerland: Site Nr. 1 - Jean-Paul Schmid, MD, ... recruiting / Virga Jesseziekenhuis,Hasselt, Belgium: Site No. 2 - Paul Dendale,MD,.... recruiting / Medical University of Gdansk, Poland, Site No. 3 - Dominika Zielinska,PhD,.... recruiting / Cliniques Universitaires Saint Luc, Brussel, Belgium: Site No. 4 - Christian Brohet,MD Prof.... recruiting / State Hospital for Cardiology, Balantonfüred, Hungary: Site No. 5 - Gabor Veress, MD Prof, ...recruiting

ELIGIBILITY:
Inclusion Criteria:

* First ICD implant within past 12 weeks
* Agrees to sign patient/partner informed consent

Exclusion Criteria:

* Angina pectoris CCS III & IV
* NYHA functional class IV
* Inability to follow rehabilitation programme
* Exercise limitations due to clinical condition
* Symptomatic exercise-induced tachyarrhythmias
* Any major non-cardiac condition that would adversely affect survival during study duration
* Unable to comply to study procedures
* Participates in a concurrent study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Study Completion 2009-12

PRIMARY OUTCOMES:
Anxiety and Depression

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Schmid, Principal Investigator — Switzerland - University Hospital (Inselspital) Bern
Locations (1):
- University Hospital (Inselspital) Berne, Bern, Switzerland